CLINICAL TRIAL: NCT07062874
Title: Combined Effect of Aerobic and Resistance Exercise in Non Ischemic Dilated Cardiomyopathy Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0359
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: CARDIOMYOPATHY
Keywords: Cardiomyopathy, Dyspnea, Exercise, Functional Independence, NIDCM.
MeSH Terms: conditions — Cardiomyopathies; Dyspnea; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined Aerobic and Resistance Exercise: (Experimental): Participants performed aerobic training three times a week for six weeks.
  Each session included a 10-minute warm-up, 30-minute main aerobic activity (60-85% of heart rate reserve using the Karvonen formula), and 10-minute cool-down.
  Additionally, they performed resistance exercises for upper and lower extremities using TheraBands, 8-10 sets covering major muscle groups, three times a week.
  Interventions: Behavioral: Combined Aerobic and Resistance Exercise; Behavioral: Aerobic Exercise Only
- Aerobic Exercise Only (Active Comparator): Participants followed the same aerobic training protocol as Group A.
  No resistance training was included.
  Sessions also occurred three times a week for six weeks, with similar warm-up, active, and cool-down phases.
  Interventions: Behavioral: Aerobic Exercise Only

INTERVENTIONS:
Behavioral: Combined Aerobic and Resistance Exercise — Participants received supervised exercise training 3 times per week for 6 weeks. Each session included a 10-minute warm-up (walking at 1.5 km/h), a 30-minute aerobic phase at 60-85% heart rate reserve (calculated using the Karvonen formula), and a 10-minute cool-down (walking at 1 km/h). In addition, participants performed resistance training for upper and lower extremities using TheraBands, with 8-10 sets targeting major muscle groups.
  Other Names: Resistance training
  Arms: Combined Aerobic and Resistance Exercise:
Behavioral: Aerobic Exercise Only — Participants followed the same aerobic training protocol as the experimental group-3 sessions per week for 6 weeks, with 10-minute warm-up, 30-minute aerobic exercise (60-85% HRR), and 10-minute cool-down. No resistance training was provided.

SUMMARY:
This study explores the effects of combined aerobic and resistance exercise in patients with non-ischemic dilated cardiomyopathy (NIDCM). In a six-week randomized clinical trial with 66 participants, both exercise groups-combined and aerobic-only-showed significant improvements in exercise capacity, functional independence, dyspnea, and blood pressure. However, no significant difference was found between the two groups. The study concludes that both exercise approaches are effective, but longer studies are needed to determine if combined training offers added benefits.

DETAILED DESCRIPTION:
The study titled "Combined Effect of Aerobic and Resistance Exercise in Non-Ischemic Dilated Cardiomyopathy Patients" by Arooj Fatima investigates how integrating both aerobic and resistance exercises impacts patients suffering from NIDCM, a condition marked by left ventricular dysfunction and reduced exercise tolerance. Through a randomized clinical trial involving 66 patients divided into two groups-one receiving both aerobic and resistance training and the other only aerobic training-the study evaluated changes in ejection fraction, VO₂ max, dyspnea, and functional independence over six weeks. Significant improvements were observed within both groups across all measured outcomes, including increased exercise capacity, better functional independence, and reduced blood pressure and dyspnea levels. However, no statistically significant difference was found between the two groups, indicating that while both exercise regimens are beneficial, the combined approach did not yield superior results within the study's timeframe. The research highlights the value of structured exercise in improving cardiovascular and functional outcomes in NIDCM patients and recommends longer, more varied studies to further explore these benefits.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female Age 40 to 60
* Left ventricular ejection fraction <50%

Exclusion Criteria:

* Patients diagnosed with valvular heart disease, supraventricular arrhythmias, congenital heart disease were excluded.
* Neuromuscular diseases such as stroke, Parkinson.
* Underlying pulmonary disease
* Impaired cognitive function (14)

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-07-28 (Estimated); Primary Completion 2025-09-28 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Functional Independence Measure (FIM) questionnaire | Baseline and 6 weeks
  Assesses level of functional independence across self-care, mobility, communication, and social cognition.
VO₂ Max (Maximum Oxygen Consumption) | Baseline and 6 weeks.
  Measured using Graded Exercise Test (GXT) to assess cardiovascular fitness.

SECONDARY OUTCOMES:
Modified Borg Dyspnea Scale | Baseline and 6 weeks.
  Rates severity of dyspnea (shortness of breath) from 0 (none) to 10 (maximum).
Blood Pressure (Systolic and Diastolic) | Baseline and 6 weeks.
  Measured via Transthoracic Echocardiogram and standard BP monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Arjumand Bano, MS-CPPT, Principal Investigator — Riphah International University
Locations (1):
- Arjumand, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No